CLINICAL TRIAL: NCT02456090
Title: PaTH Clinical Data Research Network (CDRN) Study of Healthy Lifestyles and Health Care
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Temple University (Other); Johns Hopkins University (Other); Penn State University (Other); Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Kathleen McTigue, Professor, University of Pittsburgh
Other Study IDs: STUDY20110295
Record Dates: First submitted 2015-05-26; First posted 2015-05-28 (Estimated); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Weight
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the PaTH Clinical Data Research Network (CDRN) Study of Healthy Lifestyles, Body Weight and Health Care is to use clinical data from electronic health records (EHR) and patient reported outcomes (PRO) to answer questions of clinical importance to patients, providers, and other stakeholders.

DETAILED DESCRIPTION:
The primary objective is to create the PaTH Clinical Data Research Network (CDRN) Study of Healthy Lifestyles, Body Weight and Health Care, which will allow the conduct of patient-centered observational studies on weight across the multiple institutions of the PaTH network. Creating the PaTH Clinical Data Research Network (CDRN) Study of Healthy Lifestyles, Body Weight and Health Care will involve:

1. Recruiting patients with longitudinal weight data in the EHR to participate in the PaTH Clinical Data Research Network (CDRN) Study of Healthy Lifestyles, Body Weight and Health Care
2. Administering surveys to the PaTH Clinical Data Research Network (CDRN) Study of Healthy Lifestyles, Body Weight and Health Care approximately every 6 months to collect patient reported outcomes (PROs)
3. Collecting individual patient health record data into the PaTH Clinical Data Research Network (CDRN) Study of Healthy Lifestyles, Body Weight and Health Care database
4. Identifying potential participants for future research studies.
5. Tracking whether the patient participant has biospecimens in a PaTH site biorepository and prepare for possible sharing of biospecimens in future studies.

The secondary objectives are to use the PaTH Clinical Data Research Network (CDRN) Study of Healthy Lifestyles, Body Weight and Health Care to answer patient-centered research questions including:

(1) How do survey response rates, sample demographics and survey responses differ by recruitment technique? (2) What are patients' weight management strategies? How much are health care providers contributing to their weight management approaches? Do these relationships vary by weight status, region, age, sex, or race; (3) What are patients' reasons for seeking bariatric surgery and expectations in terms of weight change?; (4) Among patients seeking bariatric surgery, what proportion with high risk for sleep apnea by survey responses have been evaluated for or diagnosed with this health problem? (5) How does physical activity vary with patients co-morbidity status?

ELIGIBILITY:
Inclusion Criteria:

* Age in years (>= 18 years), at the time of the initial data query
* Height - at least 1 at any time; can be outside 5-year cohort time window
* Weight : Two encounters each with weight within the 5-year cohort time window

Exclusion Criteria:

* Deceased
* Not proficient in English
* Already enrolled in the PaTH Clinical Data Research Network (CDRN) Study of Healthy Lifestyles, Body Weight and Health Care in another PaTH institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential participants for the PaTH Clinical Data Research Network (CDRN) Study of Healthy Lifestyles, Body Weight and Health Care will include patients identified through EHRs at the participating PaTH sites, using the eligibility criteria defined through the PCORnet Obesity Task Force and described below. We aim to recruit as many patients as possible from the target population, with one of the recruitment strategies producing a 50% enrollment rate.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2015-05; Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Create PaTH Clinical Data Research Network (CDRN) Study of Healthy Lifestyles, Body Weight and Health Care | 18 months
  Create the PaTH Clinical Data Research Network (CDRN) Study of Healthy Lifestyles, Body Weight and Health Care, which will allow the conduct of patient-centered observational studies on weight across the multiple institutions (Hershey Penn State, University of Pittsburgh, Temple University) of the PaTH network.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen McTigue, MD, Principal Investigator — University of Pittsburgh
Locations (5):
- United States (5):
  - Johns Hopkins University, Baltimore, Maryland
  - Geisinger, Danville, Pennsylvania
  - Jody McCullough, Hershey, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Bramante CT, McTigue KM, Lehmann HP, Clark JM, Rothenberger S, Kraschnewski J, Lent MR, Herring SJ, Conroy MB, McCullough J, Bennett WL. Understanding Primary Care Patients' Self-weighing Habits: Cohort Analysis from the PaTH Clinical Data Research Network. J Gen Intern Med. 2019 Sep;34(9):1775-1781. doi: 10.1007/s11606-019-05153-w. Epub 2019 Jul 16. PMID 31313111
- [Background] Jain S, Rothenberger SD, Bennett WL, Clark JM, Conroy MB, Herring SJ, Kraschnewski JL, Lent MR, Bramante CT, Cappella N, McTigue KM. Provider Advice and Patient Perceptions on Weight Across Five Health Systems. Am J Prev Med. 2020 Sep;59(3):e105-e114. doi: 10.1016/j.amepre.2020.03.013. Epub 2020 May 21. PMID 32446748
- [Background] Bennett WL, Bramante CT, Rothenberger SD, Kraschnewski JL, Herring SJ, Lent MR, Clark JM, Conroy MB, Lehmann H, Cappella N, Gauvey-Kern M, McCullough J, McTigue KM. Patient Recruitment Into a Multicenter Clinical Cohort Linking Electronic Health Records From 5 Health Systems: Cross-sectional Analysis. J Med Internet Res. 2021 May 27;23(5):e24003. doi: 10.2196/24003. PMID 34042604